CLINICAL TRIAL: NCT00526734
Title: A Randomised, International, Open-label, Phase II Study of Peripheral Blood Progenitor Cell (PBPC) Mobilization and Engraftment With Pegfilgrastim or Filgrastim for Autologous Transplantation in Patients With Multiple Myeloma (MM)
Brief Title: High-Dose Chemotherapy and Stem Cell Transplant in Treating Patients With Newly Diagnosed Stage I, Stage II, or Stage III Multiple Myeloma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasme University Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: ERA-2006-001; CDR0000561733 (Registry Identifier: PDQ (Physician Data Query)); ERA-NEUMOBIL; EUDRACT-2006-000891-34
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2007-09

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Filgrastim; pegfilgrastim; Melphalan

INTERVENTIONS:
Biological: filgrastim
Biological: pegfilgrastim
Drug: melphalan
Procedure: autologous hematopoietic stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as melphalan, use different ways to stop cancer cells from dividing so they stop growing or die. Stem cell transplant using stem cells from the patient may be able to replace immune cells that were destroyed by chemotherapy used to kill cancer cells. Giving colony-stimulating factors, such as G-CSF or pegfilgrastim, helps stem cells move from the bone marrow to the blood so they can be collected. It is not yet known which regimen is more effective in treating multiple myeloma.

PURPOSE: This randomized phase II trial is studying how well high-dose chemotherapy followed by stem cell transplant works in treating patients with newly diagnosed stage I, stage II, or stage III multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare engraftment of peripheral blood progenitor cells (PBPCs) mobilized by 2 different fixed doses of pegfilgrastim versus a by-weight dose of filgrastim (G-CSF).

Secondary

* Determine the ability of 2 different fixed doses of pegfilgrastim to mobilize PBPCs.
* Determine the safety of pegfilgrastim during PBPC mobilization and collection.
* Determine the effect of different induction chemotherapy regimens on autologous progenitor cell transplantation.

OUTLINE: This is a multicenter study. Patients are stratified by type of induction chemotherapy (Thal/Dex vs VAD vs Vel-Dex vs VTD) and by stage of disease according to International Prognostic Index criteria (stage I [i.e., beta-2 microglobulin < 3.5 and albumin > 35] vs stages II and III).

* Induction therapy: Patients receive 3-4 courses of 1 of the following regimens:

  * VAD: Patients receive vincristine, doxorubicin hydrochloride, and dexamethasone.
  * Thal/Dex: Patients receive thalidomide and dexamethasone.
  * Vel-Dex: Patients receive bortezomib and dexamethasone.
  * VTD: Patients receive bortezomib, thalidomide, and dexamethasone. Patients achieving complete, partial, or minimal response after 3-4 courses of induction therapy proceed to peripheral blood progenitor cell (PBPC) mobilization 17 days after completion of induction therapy.
* PBPC mobilization: Patients are randomized to 1 of 3 arms.

  * Arm I: Patients receive filgrastim subcutaneously (SC) once daily until the final leukapheresis.
  * Arm II: Patients receive a single dose of pegfilgrastim SC.
  * Arm III: Patients receive pegfilgrastim as in arm II at a higher dose.
* Leukapheresis: Patients undergo up to 3 leukaphereses to obtain adequate numbers of CD34-positive filgrastim- or pegfilgrastim-mobilized PBPCs for engraftment. Patients achieving a sufficient number of collected PBSCs proceed to conditioning chemotherapy.
* Conditioning chemotherapy: Patients receive high-dose melphalan* IV over 1-2 days. Patients then proceed to PBPC transplantation.

NOTE: *Patients ≥ 65 years old receive melphalan at a lower dose.

* Autologous PBPC transplantation: Patients undergo infusion of PBPCs on day 0. Patients in all arms receive G-CSF support beginning on day 1 after PBPC transplantation and continuing until blood counts recover for 3 consecutive days.

After completion of study therapy, patients are followed for up to 100 days post-transplantation.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of symptomatic stage I or stage II-III multiple myeloma

  * Newly diagnosed disease
* No amyloidosis

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-2
* ANC ≥ 1.0 x 10^9/L (without colony-stimulating factors)
* Platelet count ≥ 50 x 10^9/L (without transfusion support within the past 7 days)
* Serum calcium < 14 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 times ULN
* Creatinine clearance ≥ 50 mL/min
* Fertile patients must use effective contraception
* Negative pregnancy test
* Willing and able to comply with protocol requirements

Exclusion criteria:

* Myocardial infarction within the past 6 months
* New York Heart Association class III or IV heart failure
* Uncontrolled angina
* Severe uncontrolled ventricular arrhythmia
* Acute ischemia or active conduction system abnormalities as evidenced by ECG
* Serious medical condition that could prolong hematological recovery or preclude completion of or tolerance to protocol therapy
* Seropositive for HIV antibody
* Known hepatitis B surface antigen positivity OR active hepatitis C infection
* Active systemic infection requiring treatment
* Pregnant or nursing
* Poor psychiatric condition

PRIOR CONCURRENT THERAPY:

* No plasmapheresis within the past 4 weeks
* No major surgery within the past 4 weeks
* No anticancer therapy within the past 5 years, except treatment for basal cell carcinoma of the skin or carcinoma in situ of the uterine cervix
* No other concurrent G-CSF growth factors
* No concurrent enrollment in another investigational clinical trial
* No concurrent investigational agent that would contraindicate the use of pegfilgrastim as either a mobilization agent or a hematological recovery agent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-02

PRIMARY OUTCOMES:
Number of patients with engraftment after induction chemotherapy

SECONDARY OUTCOMES:
Number and proportion of patients from whom ≥ 2 x 10e6 CD34-positive cells/kg are harvested
Number and proportion of patients from whom ≥ 4 x 10e6 CD34-positive cells/kg are harvested
CD34-positive cells/kg yield in each leukapheresis
Number of leukaphereses to collect ≥ 2 x 10e6 CD34-positive cells/kg
Number of leukaphereses to collect ≥ 4 x 10e6 CD34-positive cells/kg
Proportion of patients with platelet recovery ≥ 20 x 10e9/L in the absence of transfusion for at least 7 days
Proportion of patients with ANC recovery of ≥ 0.5 x 10e9/L
Time to neutrophil recovery, defined as the time to neutrophil engraftment (i.e., ANC ≥ 0.5 x 10e9/L for 3 consecutive days)
Time to ANC ≥ 1.0 x 10e9/L
Time to platelet recovery, defined as the time to platelets ≥ 20 x 10e9/L in the absence of platelet transfusion support for at least 7 days
Incidence and duration of hospitalization during mobilization phase and during post-transplantation phase
Incidence and severity of adverse events during and after the use of pegfilgrastim 12 mg or pegfilgrastim 18 mg and filgrastim

CONTACTS AND LOCATIONS:
Overall Officials: Walter Feremans, MD, PhD, Study Chair — Erasme University Hospital
Locations (4):
- Hopital Universitaire Erasme, Brussels, Belgium
- Poland (3):
  - Medical University of Gdansk, Gdansk
  - Silesian Medical Academy, Katowice
  - Institute of Haematology and Blood Transfusion, Warsaw